CLINICAL TRIAL: NCT04748809
Title: An Evaluator-blinded Randomized Controlled Trial Study of the Effect of Anti-inflammatory Diet in Subjects With Rheumatoid Arthritis.
Brief Title: Effect of Anti-inflammatory Diet in Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Monica Guma, Associate Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 191900
Record Dates: First submitted 2021-01-26; First posted 2021-02-10 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm_1 (Active Comparator): Anti-inflammatory diet 1
  Interventions: Other: Diet 1
- Arm_2 (Experimental): Anti-Inflammatory diet 2
  Interventions: Other: Diet 2

INTERVENTIONS:
Other: Diet 1 — Dietary intervention
  Other Names: anti-inflammatory diet 1
  Arms: Arm_1
Other: Diet 2 — Dietary intervention
  Other Names: anti-inflammatory diet 2
  Arms: Arm_2

SUMMARY:
In a previous exploratory study, the investigators observed an effect on disease activity outcomes of anti-inflammatory diet. The investigators also observed change in microbiome and circulating metabolites. The current study will determine whether or not the addition of anti-inflammatory diet improves the clinical outcomes in participants with rheumatoid arthritis, and the role of microbiome and circulating metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low or moderate disease activity (defined as Clinical Disease Activity Index ≤ 22) and without changes in disease activity or therapy during the previous 3 months, who are interested in dietary intervention, and are able to provide consent and attend to follow up visits.

Exclusion Criteria:

* Pregnancy or lactating. Patients that will become pregnant during the study will be remove from the study.
* Food allergies
* Subjects with significant other comorbidities and /or medication use which in physician's clinical judgment might difficult the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Decrease of more than 5 points in Clinical Disease Activity Index | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No